CLINICAL TRIAL: NCT06093984
Title: A Randomized Clinical Trial Comparing Cumulative Live Birth Rates in Dual Ovarian Stimulation Versus Two Antagonist Stimulations in Poor Ovarian Responders
Brief Title: Cumulative Live Birth Rates in Dual Ovarian Stimulation Versus Two Antagonist Stimulations in Poor Ovarian Responders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: shanghaiFMIH-20231006
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Stimulation Protocol (Experimental): Dual stimulations were performed during the follicular and luteal phases in the same cycle.
  Interventions: Procedure: duostim vs. two antagonist ovarian stimulations
- Antagonist Stimulation Protocol (Active Comparator): Antagonist stimulations were performed during two consecutive follicular phases in two cycles.
  Interventions: Procedure: duostim vs. two antagonist ovarian stimulations

INTERVENTIONS:
Procedure: duostim vs. two antagonist ovarian stimulations — Human menopausal gonadotropin (HMG) 300 IU/day with flexible antagonist protocol is used for ovarian stimulation, except in luteal phase stimulation of the duostim group. In the duostim group, all of the embryos are frozen. Fresh transfers are performed in the control group, frozen embryo transfers are performed in both control and duostim groups.

SUMMARY:
To compare the difference in cumulative live birth rates between dual ovarian stimulation and two antagonist stimulations in poor ovarian responders.

DETAILED DESCRIPTION:
Studies have shown the ability to obtain oocytes with equivalent quality from the follicular and the luteal phase, and a higher number of oocytes within one cycle when using dual ovarian stimulation (duostim). This could be particularly relevant for women with poor ovarian responders (POR). Whether the cumulative live birth rates differ after duostim and two antagonist stimulations in POR remains controversial.

ELIGIBILITY:
Inclusion Criteria:

* Women with POR were defined with adjusted Bologna criteria, at least two of the three following criteria: advanced maternal age (40 years); 3 oocytes in previous IVF; and antral follicle count (AFC) 5 and/or anti-Mu¨llerian hormone (AMH) 1.1 ng/ml (this criterion was mandatory)
* Aged from 20 to 44 years
* Body mass index (BMI) from 19 to 32 kg/m2
* No more than two previous IVF cycles were recruited

Exclusion Criteria:

* Amenorrhoea
* Follicle stimulating hormone (FSH) 20 IU/L or AFC 1
* Women with a partner with an extremely severe sperm anomaly or sperm donor use

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate | 36 months
  Live birth is defined as the delivery of any alive infant after 22 weeks of gestation after our interventions, and cumulative live birth rate is calculated by the total number of women randomized to the specific group.

SECONDARY OUTCOMES:
Time to live birth (TTLB) | 36 months
  The TTLB was measured as the time from ovarian stimulation to a live birth.
Total amount of Gn used during ovarian stimulation | 24 months
  Total amount of Gn used during ovarian stimulation
Number of retrieved oocytes | 24 months
  Number of retrieved oocytes after ovarian stimulation.
Clinical pregnancy rate | 36 months
  Twenty days after conception, transvaginal ultrasonography will be performed. Clinical pregnancy will be diagnosed with detection of an intrauterine gestational sac.